CLINICAL TRIAL: NCT05315778
Title: Anti-BCMA CAR T-Cell Therapy for Relapsed/Refractory Immune Thrombocytopenia
Brief Title: Anti-BCMA CAR T-Cell Therapy for R/R ITP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCRITP
Record Dates: First submitted 2022-03-31; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: ITP
Keywords: CAR-T; BCMA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-BCMA CAR T-cells infusion (Experimental): R/R ITP patients will accept infusion of autologous anti-BCMA CAR T-cells with a total of 1.0-2.0×10e7/Kg. The patients will be follow-up for 6 months post CAR T-cell therapy.
  Interventions: Biological: autologous anti-BCMA chimeric antigen receptor T cells

INTERVENTIONS:
Biological: autologous anti-BCMA chimeric antigen receptor T cells — Lymphoadenodepletion chemotherapy with FC (fludarabine 30mg/ m2 for 3 consecutive days and cyclophosphamide 300mg/m2 for 3 consecutive days) will be given at day -5, -4 and -3 before CAR T-cells infusion. A total of 1.0-2.0×10e7/Kg autologous anti-BCMA CAR T-cells will be infused by dose-escalation after the lymphoadenodepletion chemotherapy. Dose of CAR T-cells are allowed to be adjusted according to the severity of cytokine release syndrome.

SUMMARY:
This is a prospective, single-center, open-label, single-arm study, to evaluate the efficacy and safety of Anti-BCMA chimeric antigen receptor T cell therapy（BCMA CAR-T）for patients with relapse/refractory Immune thrombocytopenia(R/R ITP).

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a disorder that can lead to easy or excessive bruising and bleeding. Approximately two-thirds of patients achieve remission after/during first-line therapies. However, the other part of patients could not achieve durable remission or even refractory to initial treatments. Those cases, known as relapse/refractory Immune thrombocytopenia (R/R ITP), undergo the heavy burden of disease which decreases the quality of life. Lots of pathogeneses take part in the occurrence of R/R ITP, and the most important one of them is antibody-mediated immune platelet destruction. As far as it is known，human platelet autoantibodies are mainly secreted by plasma cells, especially long-lived plasma cells. Researchers want to explore that can BCMA CAR-T help R/R ITP patients increase platelet count, reduce bleeding episodes and the dose of concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Refractory ITP defined according to the recent consensual criteria ( 'Chinese guideline on the diagnosis and management of adult primary immune thrombocytopenia (version 2020)'), or relapse ITP defined as ITP patients who have responded to first-line therapy (glucocorticoids or immunoglobulins) and anti-CD20 monoclonal antibody, but cannot maintain the response.
* Ages 18-65 years inclusive.
* Adequate venous access for apheresis or venous blood and no other contraindications for leukocytosis.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Subjects should have full capacity for civil conduct, understand necessary information，sign the informed consent form voluntarily，and have good corporation with the content of this research protocol.

Exclusion Criteria:

* Secondary ITP.
* Patients with a known history or prior diagnosis of arterial thrombosis (such as cerebral thrombosis, myocardial infarction, etc.), or comorbidity of venous thrombosis (such as deep vein thrombosis, pulmonary embolism), or are using anticoagulant/antiplatelet drug at the beginning of trial.
* Patients with a known history or prior diagnosis of serious cardiovascular disease.
* Patients with uncontrolled infection, organ dysfunction or any uncontrolled active medical disorder that would preclude participation as outlined.
* Patients with malignancy or history of malignancy.
* Failed T cell expansion test.
* During screening, hemoglobin <100g/L; absolute value of neutrophil count <1.5×10^9/L.
* During screening, serum creatinine concentration > 1.5x the upper limit of the normal range, total bilirubin > 1.5x the upper limit of the normal range, alanine aminotransferase and aspartate aminotransferase > 3x the upper limit of the normal range, Left ventricular ejection fraction ≤ 50% by echocardiography, Pulmonary function ≥ grade 1 dyspnea (CTCAE v5.0), blood oxygen saturation<91% without oxygen inhalation.
* Prothrombin time (PT) or prothrombin time-international normalized ratio (PT-INR) or activated partial thromboplastin time (APTT) exceeding 20% of the normal reference range; or a history of coagulation abnormalities other than ITP.
* Either HIV antibody or syphilis antibody is positive; hepatitis C antibody is positive and the detection of HCV-RNA exceeds the laboratory test upper reference limit; hepatitis B surface antigen is positive and the detection of HBV-DNA exceeds the laboratory test upper reference limit.
* Participated in other clinical studies within 3 months before this CAR-T cell infusion.
* Patients is pregnant or breastfeeding, or planning pregnancy.
* Patients is fertile and the investigator determines the case is inappropriate to participate.
* History of severe drug allergy or known allergy to CAR-T treatment related drugs.
* Suspected or established alcohol, drug or drug abuse.
* The investigator judges that it is not suitable to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
overall response | 6-months
  The number of participants who achieved CR (defined as platelet count≥100x10e9/L) and PR (defined as platelet count ≥30x10e9/L and at least a 2-fold increase the baseline count and absence of bleeding) at follow-up.

SECONDARY OUTCOMES:
Time to response | 6-months
  Time since infusion of CAR T-cells to the time to achieve the response.
Duration of response | 6-months
  Period from the achievement of response to the loss of response.
Incidence of adverse events | 6-months
  Adverse events will be assessed daily during the first 2 weeks after the BCMA CAR-T treatment, and monthly thereafter. Adverse events will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Evaluation of bleeding events | 6-months
  Bleeding events will be evaluated according to Bleeding rating system of ITP('Chinese guideline on the diagnosis and management of adult primary immune thrombocytopenia (version 2020)').
Evaluation of concomitant therapy | 6-months
  Duration of discontinuation or dose reduction of concomitant treatment，and the degree of decrease of combined treatment from the baseline in patients.
Evaluation of health-related quality of life | 6-months
  Health-related quality of life will be evaluated according to ITP-PAQ (Primary Immune Thrombocytopenia Patient Assessment Questionnaire).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided